CLINICAL TRIAL: NCT01798472
Title: Cemented Versus Uncemented Arthroplasty in Elderly Patients With Displaced Femoral Neck Fractures: a Randomized Controlled Trial
Brief Title: Hip Fractures Treated With Uncemented Arthroplasties
Acronym: HUA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stockholm South General Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Inngul, Consultant orthopeadic surgery, Stockholm South General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1188-31/1
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Femoral Neck Fractures
Keywords: displaced femoral neck fractures; treatment; uncemented arthroplasty; cemented arthroplasty
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Bone Cements; Cimetidine; Marathon Running

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- uncemented hemiarthroplasty (Experimental): Patients aged 80 or older with displaced femoral neck fracture treated with an uncemented hemiarthroplasty
  Interventions: Procedure: uncemented hemiarthroplasty
- reverse hybrid total hip arthroplasty (Experimental): Patients aged between 65 and 79 years treated with an reverse hybrid arthroplasty.
  Interventions: Procedure: reverse hybrid total hip arthroplasty
- cemented hemiarthroplasty (Active Comparator): Patients aged 80 or older with displaced femoral neck fracture treated with an cemented hemiarthroplasty
  Interventions: Procedure: cemented hemiarthroplasty
- cemented total hip arthroplasty (Active Comparator): Patients aged between 65 and 79 years treated with an cemented total hip arthroplasty.
  Interventions: Procedure: cemented total hip arthroplasty

INTERVENTIONS:
Procedure: cemented hemiarthroplasty — Patients aged 80 years and older operated with an cemented hemiarthroplasty. Fixation of the wedge-shaped, polished ChromCobalt steel femoral stem to host bone by use of PolyMetylMetAcrylat bone cement. The acetabulum is not replaced. The prosthesis articulates with the patients acetabulum with an unipolar, femoral head made of ChromCobalt steel.
  Other Names: Femoral stem, Exeter, Stryker; Unipolar femoral head, Stryker; Bone cement, Optipac, Biomet
  Arms: cemented hemiarthroplasty
Procedure: reverse hybrid total hip arthroplasty — Patients aged 65 to 79 years operated with an uncemented femoral component combined with cemented acetabular cup. The femoral stem is fixed to the host bone by press-fit technique. We use a tapered, proximally hydroxyapatite coated, titanium stem. The acetabular cup is fixed to the host bone with bone cement. We use an all-polyethylene design. Bone cement consists of PolyMetylMetAcrylat.
  Other Names: Femoral stem: Bimetric, Biomet; Acetabular cup, Maraton, DePuy; Bone cement, Optipac, Biomet
  Arms: reverse hybrid total hip arthroplasty
Procedure: cemented total hip arthroplasty — Patients aged 65 to 79 years operated with a cemented femoral stem combined with a cemented acetabular cup. Femoral and acetabular component are fixed to the host bone by use of bone cement. The femoral stem is a polished, wedge-shaped design made of ChromCobalt steel. The acetabular cup is fixed to the host bone with bone cement.The acetabular cup an all-polyethylene design. Bone cement consists of PolyMetAcrylat.
  Other Names: Femoral stem: Exeter, Stryker; Acetabular cup, Marathon, DePuy; Bone cement, Optipac, Biomet
  Arms: cemented total hip arthroplasty
Procedure: uncemented hemiarthroplasty — Patients aged 80 years and older are randomized to uncemented hemiarthroplasty. Fixation of the tapered, proximally hydroxyapatite coated, titanium stem to the host bone by "press-fit"-technique. The acetabulum is not replaced. The prosthesis articulates with the patients acetabulum with an unipolar, femoral head made of ChromCobalt steel.
  Other Names: Femoral stem: Bimetric, Biomet; Femoral head: Biomet
  Arms: uncemented hemiarthroplasty

SUMMARY:
The aim of this study is to compare the functional and radiological outcome after displaced, femoral neck fractures treated with either cemented or uncemented arthroplasties.

The primary hypothesis is that the uncemented arthroplasty shows the same functional outcome at 12 month as the cemented arthroplasty.

DETAILED DESCRIPTION:
Femoral neck fracture is a common cause of suffering and premature mortality among the elderly. Riskfactors for femoral neck fractures are age, gender, osteoporosis and cognitive dysfunction.

Mortality and morbidity varies between undisplaced and displaced femoral neck fractures.

Different treatment options are available: reduction and internal fixation vs joint replacement (arthroplasty). The treatment of undisplaced femoral neck fractures is uncontroversial and consists of internal fixation with screws.

The treatment of displaced, femoral neck fractures with internal fixation shows unacceptable results with complications rates leading to reoperation between 40-60%. Treatment of these fractures with arthroplasties has therefore become the standard treatment in industrial countries.

Fixation of the femoral component with bone-cement is standard procedure in Europe today. To avoid negative cardio-pulmonary events in patients with serious comorbidities and in very old and frail patients uncemented femoral components or internal fixation are used. These uncemented stems are mostly older design with poor track records. The use of modern, well-documented stems used in an osteoarthritis population for fracture patients has still to be tested.

ELIGIBILITY:
Inclusion Criteria:

* displaced fracture of the femoral neck
* independent living
* independent ambulation (with or without walking aids)

Exclusion Criteria:

* pathological fracture
* severe dementia (defined as ≤3 in short portable mental questionnaire) preoperatively
* preexisting ipsilateral hip disease
* neurological disease (e.g. M. Parkinson)
* psychiatric disease which makes understanding or following instructions impossible
* history of drug and alcohol abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-11; Primary Completion 2016-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 12 month
  Our primary outcome variable is the Harris Hip Score at 12 month follow up. Harris Hip Score is an investigator reported tool evaluating hip function in four dimensions:
  Pain, function, absence of deformity and range of motion

SECONDARY OUTCOMES:
Health related quality of life | 12 month
  We use the patient reported instrument EQ-5D. A questionnaire consisting of 5 questions to evaluate health related quality of life.
Radiological follow up | 12 month
  Evaluation of radiological outcome on standard hip radiographies with focus on bony ingrowth, signs of loosening and subsidence

OTHER OUTCOMES:
General and surgical complications | from operation until 12 month postoperatively
  general complications such as cardio-pulmonary events, pressure ulcer, pneumonia, deep vein thrombosis (DVT).
  surgical complications such as infections, reoperations due to all causes, dislocations

CONTACTS AND LOCATIONS:
Overall Officials: Sari Ponzer, M.D. Prof, Study Director — Department of orthopedic surgery, South general hospital, Sjukhusbacken 10, 118 83 Stockholm, Sweden
Locations (1):
- Södersjukhuset (South general hospital), Department of orthopedic surgery, Stockholm, Sweden